CLINICAL TRIAL: NCT03377465
Title: Biomarkers, Hemodynamic and Echocardiographic Predictors of Ischemic Strokes and Their Influence on the Course and Prognosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Paulina Gąsiorek, Principal Investigator, Medical University of Lodz
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01122017
Record Dates: First submitted 2017-12-05; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Embolic Stroke of Undetermined Source; Ischemic Stroke; Atrial Fibrillation and Flutter; Myocardial Infarction; Cardiac Tumor; Endocarditis; Patent Foramen Ovale
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Myocardial Infarction; Heart Neoplasms; Endocarditis; Foramen Ovale, Patent

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients with stroke of undetermined cause age 18-65
  Interventions: Diagnostic Test: ADMA (asymmetric dimethylarginine) , NTproBNP (N-terminal pro b-type natriuretic peptide), IL-6 (Interleukin 6), Adiponectina, Leptine, Syndecan, Resistin
- Comparative group (Active Comparator): Healthy patients age 18-65
  Interventions: Diagnostic Test: ADMA (asymmetric dimethylarginine) , NTproBNP (N-terminal pro b-type natriuretic peptide), IL-6 (Interleukin 6), Adiponectina, Leptine, Syndecan, Resistin

INTERVENTIONS:
Diagnostic Test: ADMA (asymmetric dimethylarginine) , NTproBNP (N-terminal pro b-type natriuretic peptide), IL-6 (Interleukin 6), Adiponectina, Leptine, Syndecan, Resistin — ADMA, NTproBNP, IL-6, Adiponectina, Leptine, Syndecan, Resistin

SUMMARY:
A stroke is the second cause of deaths after heart attack, one of the most important causes of malfunction as far as adults are concerned and the second as for the frequency cause of dementia. In spite of a possibility of the therapy of stroke ( tissue plasminogen activator) and recognized most of risk factors there is expected that incidence rate on stroke connected with ageing of the society will be growing. It will cause medical and social consequences.

There are many of potential causes of cardiac strokes, which are not entirely examined.

More over many cryptogenic strokes are presumed to have an embolic etiology, and the frequent cause of these kind of strokes at young age is probably the mechanism of paradoxical embolism through patent foramen ovale.

As far as the investigators are concerned, at present there is lack of any recommendations for these scientific hypothesis.

DETAILED DESCRIPTION:
A stroke is the second cause of deaths after heart attack, one of the most important causes of malfunction as far as adults are concerned and the second as for the frequency cause of dementia. In spite of a possibility of the therapy of stroke ( tissue plasminogen activator) and recognized most of risk factors there is expected that incidence rate on stroke connected with ageing of the society will be growing. It will cause medical and social consequences.

The risk factors of stroke can be divided into alterable and not alterable. Importantly, the not alterable factors are: age, sex, race and genetic factors. After the age of 55 the risk of stroke grows twice in every decade of life. Moreover, it was alleged that incidence rate on stroke is more frequent at women than at men. At the black race the incidence rate on stroke is twice more frequent than at white race.

Well- known are also genetic syndromes connected with strokes like s. MELAS or CADASIL.

Well- known alterable factors are:

* hypertension
* coronary disease
* atrial fibrillation
* hypercholesterolemia
* diabetes
* nicotinism
* blood clotting disorder
* alcoholism
* TIA (transient ischemic attack) or previous former stroke
* asymptomatic stenosis of internal carotid artery

Cardiogenic stroke is a stroke caused by embolic material, which was created in cardiac cavities or on cardiac valves. They comprised 11% of all strokes and 25% of ischemic strokes. Additionally, among patients over 80 years old cardiac causes are responsible for even 40% of all ischemic strokes and half of cardiogenic strokes is caused of atrial fibrillation. Among young people (below 45 years old) about 50% of strokes are cardiogenic and are connected with paradoxical embolism at patients with patent foramen ovale.

Furthermore, cardiac- brain embolism is a result of:

* structural defect of cavities and valves of heart
* arrhythmia
* disturbances of movability of walls of the heart and function of endocardium which leads to increased risk of the risk of parietal thrombus
* cardiac insufficiency

There are many of potential causes of cardiac strokes, which are not entirely examined as for example:

* small pockets of intra- atrial septum
* structures in dextral atrium like Eustachian valve or Chiari network
* there is also a theory that even enlargement of left atrium may be the cause of brain stroke
* aneurysm of intra- atrial septum.

As far as the investigators are concerned, at present there is lack of any recommendations for these scientific hypothesis.

Available data suggest that in the comparison with atherosclerosis and lacunar strokes cardiogenic strokes characterize with high mortality ranging of 27%. Also the risk of relapse is higher than in strokes of other etiology.

Nevertheless, unfortunately, in spite of wide diagnostics at about 25-30% of patients with ischemic stroke the cause is unknown. This kind of stroke is called cryptogenic stroke or stroke with undefined etiology.

They constitute almost half of all ischemic stroke at young patients (below 55 years old). Many cryptogenic strokes are presumed to have an embolic etiology, and the frequent cause of these kind of strokes at young age is probably the mechanism of paradoxical embolism through patent foramen ovale.

To conclude, currently there aren't researches defining recommendations for long- lasting treatment patients with rare causes of strokes.

ELIGIBILITY:
Inclusion Criteria:

* stroke of undetermined cause

Exclusion Criteria:

* unstable hypertension
* atrial fibrillation
* hyperthyroidism hard
* pregnancy and breastfeeding
* dialysis
* cancer
* autoimmunologic disease
* active infection
* incapable of giving agreement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
physiological parameter | 24 months
  CRP (C reactive protein)
physiological parameter | 24 months
  IL-6 (interleukin 6)
physiological parameter | 24 months
  ADMA (asymmetric dimethylarginine)
physiological parameter | 24 months
  NTproB (N-terminal pro b-type natriuretic peptide)
physiological parameter | 24 months
  Adiponectin
physiological parameter | 24 months
  Leptine
physiological parameter | 24 months
  Resistin
physiological parameter | 24 months
  Syndecan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gasiorek P, Sakowicz A, Banach M, von Haehling S, Bielecka-Dabrowa A. Arterial Stiffness and Indices of Left Ventricular Diastolic Dysfunction in Patients with Embolic Stroke of Undetermined Etiology. Dis Markers. 2019 Sep 12;2019:9636197. doi: 10.1155/2019/9636197. eCollection 2019. PMID 31612072